## STATISTICAL ANALYSIS PLAN

Project Title: Barbershop Talk: HIV Prevention for African American Heterosexual Men

NCT Number: NCT01980771

Date of document: 8/16/18

To describe study sample characteristics across groups at baseline and follow-up and in relation to condomless sex, the  $\chi 2$  test for categorical variables and the independent samples t-test for group differences in continuous variables were utilized. From the original list of measured variables, only those covariates that were associated at p < 0.05 with baseline report of condomless sex or on which there were imbalances between the BTWB intervention and control groups at baseline, were included. Generalized mixed-effects models were used to estimate between-group differences at the participant level, taking into account the hierarchical data structure, with men clustered by barbershop. Differences between the BTWB intervention and control groups in changes in the outcomes were analyzed on an intention-to-treat basis. A binary logistic regression model was used to examine changes in condomless sex, with the six-month value modelled as the outcome and experimental group as the predictor, while controlling for barbershop site of recruitment (random effect), the baseline value of condom use (fixed effect), and covariates (fixed effects). Interaction terms between the covariates and experimental group assignment were tested for statistical significance in a stepwise approach. Data were analyzed using SAS PROC GLIMMIX, version 9.4, 2013.